CLINICAL TRIAL: NCT04747054
Title: Randomized Trial of Loco-regional Radiotherapy Added to Pembrolizumab Alone or With Chemotherapy Versus Systemic Treatment Alone for Patients With Newly Diagnosed Head and Neck Squamous Cell Carcinoma With Synchronous Metastases
Brief Title: Study on the Efficacy of Treatment by Radiotherapy and Pembrolizumab in Newly Diagnosed Metastatic Head & Neck Cancers
Acronym: PembroMetaRT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: GORTEC (Other); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-HNG-2007; 2020-A02221-38 (Other: ANSM)
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Metastatic; Radiotherapy; pembrolizumab; Squamous Cell Carcinoma; Head and Neck; Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Carcinoma, Squamous Cell; Carcinoma | interventions — pembrolizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy added to systemic treatment (Experimental): Pembrolizumab 200mg every 3 weeks until disease progression or unacceptable toxicity.
  Loco-regional radiotherapy(RT) depending on the RT timing :
  * Before 3 cycles of pembrolizumab: RT could start at any time between one week after the first administration of pembrolizumab and the first day of the 3rd cycle.
  * After 3 cycles of pembrolizumab: RT could start at any time after 3rd cycle and up to a maximum of 4 weeks after the 6th cycle of pembrolizumab.
  If the investigator decides before randomization to add chemotherapy and depending on the RT timing:
  * Start of RT planned before 3rd cycle: Chemotherapy could be delayed after the end of RT and start from cycle 3 or 4 of pembrolizumab.
  * RT planned after 3rd cycle: Chemotherapy should start at the same time of pembrolizumab.
  Chemotherapy will be composed of carboplatin AUC 5 mg/mL/min or cisplatin 100 mg/m² every 3 weeks with 5-fluorouracil (5-FU) 1000mg/m²/day during 4 days every 3 weeks for a maximum of 6 cycles
  Interventions: Drug: Pembrolizumab; Radiation: Loco-regional radiotherapy; Drug: Chemotherapy
- Systemic treatment (Active Comparator): Pembrolizumab 200 mg every 3 weeks until disease progression or unacceptable toxicity.
  If the investigator decides before randomization to add chemotherapy with pembrolizumab, the chemotherapy will be composed of carboplatin area under the curve (AUC) 5 mg/mL/min or cisplatin 100 mg/m² every 3 weeks with 5-FU 1000 mg/m²/day during 4 days every 3 weeks for a maximum of 6 cycles
  Interventions: Drug: Pembrolizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg every 3 weeks until disease progression (as confirmed according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1)) or unacceptable toxicity. The treatment of pembrolizumab should not be delayed because of radiotherapy planning.
  Other Names: KEYTRUDA
Radiation: Loco-regional radiotherapy — Depending on the choice of radiotherapy timing:
  * Before 3 cycles of pembrolizumab with or without chemotherapy : radiotherapy could start at any time between one week after the first administration of pembrolizumab and the first day of the 3rd cycle.
  * After 3 cycles of pembrolizumab with or without chemotherapy : radiotherapy could start at any time after 3rd cycle (C3D1) and up to a maximum of 4 weeks after the 6th cycle of pembrolizumab.
  Dose/fraction of radiotherapy: 54 Gy/18 fractions (recommended schedule) or 70Gy/33-35 fractions or other curative dose/fraction schedules with shorter duration and biologically equivalent dose of at least 60Gy at the discretion of local investigators, in the head and neck region. The volume of RT will include only involved loco-regional tumor region and no prophylactic neck volume will be necessary. Other cycles of pembrolizumab will be administered during and after radiotherapy.
  Arms: Radiotherapy added to systemic treatment
Drug: Chemotherapy — If the investigator decide to add chemotherapy with pembrolizumab, and depending on the radiotherapy timing:
  * Start of radiotherapy planned before 3rd cycle: Chemotherapy could be delayed after the end of radiotherapy and start from cycle 3 or 4 of pembrolizumab. Administration of chemotherapy can be delayed in case of non resolved grade 3 or higher toxicity from radiotherapy.
  * Radiotherapy planned after 3rd cycle: Chemotherapy should start at the same time of pembrolizumab.
  Chemotherapy will combine carboplatin AUC 5mg/mL/min or cisplatin 100mg/m² every 3 weeks with 5-FU 1000mg/m²/j during 4 days every 3 weeks for a maximum of 6 cycles

SUMMARY:
Study to evaluate the efficacy of treatment by radiotherapy and pembrolizumab in newly diagnosed metastatic head & neck cancers

DETAILED DESCRIPTION:
Comparative interventional prospective phase 3, randomised, open-label, multicentric trial comparing the combination of radiotherapy and pembrolizumab alone or with chemotherapy to systemic treatment as first line treatment of patients with newly diagnosed head and neck squamous cell carcinoma with synchronous metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent form prior to any study specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.
2. Histologically confirmed squamous cell carcinoma of head and neck (oral cavity, oropharynx, hypopharynx, and larynx) including unknown primary head and neck lymph nodes with distant metastases at presentation (T1-4 N0-3 M1). Histological confirmation is required in case of a single metastatic lesion.
3. Eligible for treatment by pembrolizumab according to the European Marketing Authorization
4. Patient ≥18 years old
5. Performance status: 0-1 (WHO)
6. Combined Positive Score (CPS) ≥1 for primary tumor (as determined per local practice)
7. Subjects must have at least one measurable lesion as per RECIST v1.1 to assess efficacy
8. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to randomization:

   a. If randomization is done before treatment start: i. Absolute neutrophil count ≥1.5 × 10⁹/L ii. Platelet ≥100 × 10⁹/L iii. Hemoglobin ≥90 g/L iv. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT), ≤3 × upper limit of normal (ULN), (unless documented liver metastases where ≤5 x ULN is permitted) v. Bilirubin ≤1.5 × ULN. vi. Serum albumin ≥25 g/L vii. Creatinine clearance ≥30 mL/min (calculated per institutional guidelines or by Cockcroft-Gault or Modification of Diet in Renal Disease (MDRD) formula) viii. Corrected serum calcium of ≤11.5 mg/dL or ≤2.6 mmol/L. b. If randomization if done after treatment start i. Absolute neutrophil count ≥1.0 × 10⁹/L ii. Platelet ≥75 × 10⁹/L iii. Hemoglobin ≥85 g/L
9. Patient must agree to use adequate contraception methods for the duration of the study treatment and up to 4 months after the last dose of pembrolizumab administration
10. Patients must be affiliated to a Social Security System (or equivalent)
11. No disease progression during systemic treatment if the randomization is done after the start of pembrolizumab for the current disease

Exclusion Criteria:

1. Symptomatic central nervous system (CNS) metastases and / or carcinomatous meningitis
2. History of another malignancy within 2 years prior to study inclusion, with the exception of completely resected basal or squamous cell skin cancer, or successfully treated in-situ carcinoma
3. Prior radiotherapy in the head and neck region
4. Any prior or current non-surgical treatment for invasive head and neck cancer. (except for pembrolizumab +/- chemotherapy for the current cancer for a maximum of 6 cycles). This will include but is not limited to: prior tyrosine kinase inhibitors, any monoclonal antibody, chemotherapy, anti-PD-1/PD-L1 and CTLA-4, prior radiotherapy (RT), or use of any investigational agent. Loco-regional recurrent or second primary head and neck cancer after prior surgical treatment alone in the head and neck region could be eligible.
5. Known Acquired Immune Deficiency Syndrome (AIDS)
6. Known currently active infection including hepatitis B or hepatitis C
7. Patient having received live attenuated vaccine within 28 days prior to enrolment
8. Pregnant or breast feeding woman
9. Active autoimmune disease except vitiligo, type-1 diabetes, hypothyroid stabilized with hormonal substitution, or psoriasis which do not require systemic treatment
10. Active immunodeficiency or ongoing immunosuppressive therapy
11. Active symptomatic interstitial lung disease
12. Significant disease which, in the judgment of the investigator, as a result of the medical interview, physical examinations, or screening investigations would make the patient inappropriate for entry into the trial
13. Any social, personal, medical, geographic and/or psychologic factor(s) that could interfere with the observance of the patient to the protocol and/or the follow-up and/or the signature of the informed consent
14. Prior organ transplantation including allogenic stem-cell transplantation
15. Other severe acute or chronic medical conditions including colitis, pneumonitis, pulmonary fibrosis or psychiatric conditions including active suicidal ideation; or laboratory abnormalities that may increase the risk associated with study participation and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
16. Person deprived of their liberty or under protective custody or guardianship
17. Patient who have taken any investigational medicinal product or have used an investigational device within 30 days prior to study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to disease progression or death, up to 3 years.
  The progression-free survival is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, up to 5 years.
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive. The outcome is to evaluate whether the radiotherapy improves overall survival compared to standard of care.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, 4 months, 6 months, 12 months, 18 months, 2 years, 3 years, and 4 years
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials. The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life Questionnaire - Head & Neck Cancer Module (QLQ-H&N35) | At baseline, 4 months, 6 months, 12 months, 18 months, 2 years, 3 years, and 4 years
  The head & neck cancer module is a 35-item questionnaire designed for use among a wide range of patients with head & neck cancer, varying in disease stage and treatment modality. It includes 7 multi-item scales that assess pain (4 items), swallowing (4 items), senses (2 items), speech (3 items), social eating (4 items), social contact (5 items), and sexuality (2 items). There are also 11 single items. Using a 4-point Likert scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), patients indicate the degree to which they have experienced symptoms. For all items and scales, high scores indicate more problems.
Objective response rate (ORR) | At 18 weeks and 27 weeks
  The Objective response rate is defined as the presence of a partial response (PR) or complete response (CR) observed at week 18 and at week 27 after randomization. The investigator will evaluate the objective response using RECIST v1.1.
Loco-regional progression | From randomization to loco-regional progression, up to 5 years.
  Locoregional disease progression is defined as the time from randomization to the first documented locoregional progression evaluated by RECIST v1.1.
Distant progression | From randomization to distant progression, up to 5 years.
  Distant progression is defined as the time from randomization to the first documented distant disease progression evaluated by RECIST v1.1.
Progression-free survival 2 (PFS2) | Up to 5 years after randomization.
  Progression-free survival 2 is defined as time from randomization to a second tumor progression (according to RECIST V1.1) on next-line treatment (given after a first progression) or death from any cause. Patients who did not have a progression after the initial treatment are counted as an event at the time of death if they died whatever the cause of death or are censored at the time of last news if they are alive. Patients who had a progression after the initial treatment are counted as an event when they progressed again under or after the treatment of the first progression (if they start a new treatment, i.e. a third treatment, they are also counted as an event) or when they died whatever the cause of death or they are censored at the time of last news if they are alive without new progression after the first progression.
Incidence of Treatment Adverse Events | Throughout study completion, up to 5 years.
  The tolerance and safety will be evaluated by toxicity (acute [<1 months after the end of pembrolizumab] and late [≥1 month after the end of pembrolizumab]), assessed using the Common terminology criteria for adverse events version 5.0 (CTCAE v5.0).
Compliance to treatment | Throughout study treatment, up to 5 years
  Compliance to treatment is defined by the difference on received study regimen compared to the planned study regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Yungan TAO, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Caroline EVEN, Dr, Principal Investigator — Gustace Roussy
Locations (26):
- France (26):
  - Institut Sainte Catherine, Avignon
  - CHU Jean Minjoz, Besançon
  - CHU Bordeaux, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - CH Carcassonne, Carcassonne
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Guillaume le Conquérant, Le Havre
  - Centre Jean Bernard - Clinique Victor Hugo, Le Mans
  - Centre Oscar Lambret, Lille
  - Groupe Hospitalier Bretagne Sud, Lorient
  - Centre Léon Bérard, Lyon
  - Hopital de la Timone, Marseille
  - Hopital Nord Franche Comté - Site de Mittan, Montbéliard
  - Centre Antoine Lacassagne, Nice
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - CHU de Saint Etienne, Saint-Priest-en-Jarez
  - Institut de Cancérologie Strasbourg-Europe, Strasbourg
  - Polyclinique de l'Ormeau, Tarbes
  - Institut Claudius Regaud, Toulouse
  - Hopital Privé Drome Ardeche, Valence
  - CH Valence, Valence
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.